CLINICAL TRIAL: NCT00088166
Title: A Phase III Randomized, Double-Blind, Dexamethasone-Sparing Study Comparing Human Corticotropin-Releasing Factor (hCRF) to Placebo for Control of Symptoms Associated With Peritumoral Brain Edema in Patients With Malignant Brain Tumor Who Require Chronic Administration of High-Dose Dexamethasone
Brief Title: XERECEPT® (hCRF) for Patients Requiring Dexamethasone to Treat Edema Associated With Brain Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celtic Pharma Development Services (Industry)
Collaborators: Neurobiological Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTI 0303; XERECEPT®; NCT00091013 (obsolete NCT alias)
Record Dates: First submitted 2004-07-20; First posted 2004-07-22 (Estimated); Results first posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-07

CONDITIONS: Brain Edema; Brain Tumor
Keywords: peritumoral brain edema; edema; malignant brain tumor; astrocytoma; brain tumor; dexamethasone; Decadron
MeSH Terms: conditions — Brain Edema; Brain Neoplasms; Edema; Astrocytoma | interventions — Corticotropin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Experimental): Patients will take hCRF (XERECEPT) 2mg/day and open label-dexamethasone they are currently taking.
  Interventions: Drug: hCRF
- II (Placebo Comparator): Patient will receive placebo hCRF and any open-label dexamethasone that they are currently taking
  Interventions: Drug: placebo hCRF

INTERVENTIONS:
Drug: hCRF — hCRF ; open-label dexamethasone that the patient is currently taking
  Other Names: XERECEPT (corticorelin acetate injection); hCRF
  Arms: I
Drug: placebo hCRF — placebo hCRF 2mg/day and open-label dexamethasone that they are taking
  Other Names: XERECEPT (corticorelin acetate injection)
  Arms: II

SUMMARY:
The purpose of this study is to compare the safety and efficacy of XERECEPT® to dexamethasone (Decadron) a common treatment for symptoms of brain swelling (edema). This study is specifically aimed at patients who require chronic high doses of dexamethasone to manage symptoms.

DETAILED DESCRIPTION:
XERECEPT® is not a potential treatment for cancer, but may reduce the edema associated with tumors and as a result, decrease neurological symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of a primary malignant brain tumor or, if metastatic, documentation and histology (if available) of primary source of cancer.
* Patient must have 1 or more qualifying steroid-associated side effect(s) at Baseline.
* Patient has required administration of dexamethasone to control symptoms of peritumoral edema for at least 30 days.
* Stable dexamethasone dose of 4-24 mg/day for at least 14 days prior to Baseline.
* Need for administration of dexamethasone to treat peritumoral brain edema (referenced above) has been documented by MRI or comparable diagnostic technology within 21 days of Baseline.
* Karnofsky score of > 50 at Screening and Baseline.
* Capable of self-administration of subcutaneous injections twice daily for 12 weeks, or availability of assistance from caregiver.
* Ability to provide written informed consent or, if unable to provide, have a legal guardian or representative provide written informed consent.
* For women of childbearing potential: a negative serum pregnancy test at Screening.
* Must be 18 years of age or older

Exclusion Criteria:

* Ongoing or anticipated need for surgery, radiosurgery or radiation therapy or the introduction of new chemotherapeutic regime within the first 5 weeks of study enrollment. Treatment with pre-study chemotherapy may continue.
* Concurrent enrollment in any other investigational drug or device study, or plan to enroll in such a study during the first 5 weeks of treatment.
* Systemic steroid use for any indication other than peritumoral brain edema.
* Use or intended use of dexamethasone as an anti-emetic during Screening or Study
* Non-compliance with dexamethasone or anticonvulsant therapy.
* Clinical signs and symptoms of cerebral herniation.
* Serious concomitant cardiovascular, pulmonary, renal, gastrointestinal or endocrine metabolic disease which could put the patient at unusual risk for study participation.
* Confounding previous or concurrent neurological disorders that would interfere with adequate clinical evaluation.
* Clinically significant head injury or chronic seizure disorder, if the condition results in functional impairment or is likely to interfere with evaluations. (Maintenance anticonvulsant therapy is allowed.)
* Central nervous system infection.
* Pregnancy, breastfeeding and/or refusal to practice birth control while in study, for women of childbearing potential.
* Any conditions that are considered contraindications for patients to receive niacin, e.g. liver disease (with LFTs > 3 times the upper limit of the norm),active peptic ulcer, arterial hemorrhage, asthma and known hypersensitivity to niacin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2004-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Shapiro, MD, Principal Investigator — Barrow Neurological Institute
Locations (34):
- United States (27):
  - Barrow Neurological Institute, Phoenix, Arizona
  - UCSF Fresno Center for Clinical Studies, Fresno, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Stanford University Medical Center, Palo Alto, California
  - UC Davis Medical Center, Division of Medical Oncology, Sacramento, California
  - UC San Diego, Thornton Hospital, San Diego, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Colorado Neurological Institute, Englewood, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - Cancer Institute of Orlando, Orlando, Florida
  - Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Hermelin Brain Tumor Center, Henry Ford Hospital, Detroit, Michigan
  - Neurology Group of Bergen County, Ridgewood, New Jersey
  - Dent Neurologic Institute, Amherst, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - University Hematology Oncology Care, LLC, Cincinnati, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oregon Clinic, Portland, Oregon
  - Virginia Mason Clinic, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (7):
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Moncton Hospital, Moncton, New Brunswick
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Kingston General Hospital, Kingston, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Sunnybrook and Women's College Health, Toronto, Ontario

REFERENCES:
- [Derived] Recht L, Mechtler LL, Wong ET, O'Connor PC, Rodda BE. Steroid-sparing effect of corticorelin acetate in peritumoral cerebral edema is associated with improvement in steroid-induced myopathy. J Clin Oncol. 2013 Mar 20;31(9):1182-7. doi: 10.1200/JCO.2012.43.9455. Epub 2013 Feb 4. PMID 23382470

RESULTS

PARTICIPANT FLOW:
Groups:
- hCRF: Patients will take hCRF (XERECEPT) 2mg/day and open label-dexamethasone they are currently taking.
- Placebo: Patient will receive placebo hCRF and any open-label dexamethasone that they are currently taking
Period: Overall Study
Arm/Group | hCRF | Placebo
Started | 100 | 100
Completed | 47 | 39
Not Completed | 53 | 61
Not completed — Adverse Event | 11 | 9
Not completed — Death | 3 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 4 | 1
Not completed — Protocol Violation | 1 | 5
Not completed — Patient deterioration | 29 | 39
Not completed — Withdrawal by Subject | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | hCRF | Placebo | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 89 | 87 | 176
  >=65 years | 11 | 13 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (11.8) | 52.7 (11.6) | 52.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 43 | 86
  Male | 57 | 57 | 114
Region of Enrollment [Number; unit: participants]
  United States | 90 | 81 | 171
  Canada | 7 | 15 | 22
  Australia | 3 | 3 | 6
  New Zealand | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients in Each Treatment Group Who Are Responders at Week 2 and Continue to be Responders at Week 5
Description: The primary efficacy endpoint was the proportion of patients in each treatment group who were Responders at Week 2 and who continued to be Responders at Week 5. Responders were defined as study patients who demonstrated the following:
  * 50% or greater reduction in dexamethasone dose relative to Baseline
  * Overall 10-Item Neurological Examination Score unchanged or lower compared to Baseline
  * Karnofsky Score unchanged or increased relative to Baseline
Time Frame: Prospective
Population: Intent to Treat Population
Measure: Number; unit: participants
Arm/Group | hCRF | Placebo
Number analyzed (Participants) | 100 | 100
participants | 57 | 46

2. Secondary Outcome: Percent of Patients in Each Treatment Group Achieving 50% Reduction in Dexamethasone Usage Relative to Baseline by Week 2 Without Deterioration in Neurological Function as Measured by the 10-Item Neurological Exam and the KPS
Time Frame: Prospective
Population: Intent to Treat Population
Measure: Number; unit: participants
Arm/Group | hCRF | Placebo
Number analyzed (Participants) | 100 | 100
participants | 78 | 62

3. Secondary Outcome: The Proportion of Patients in Each Treatment Group Who Are Responders at Week 2 and Who Continue to be Responders at Weeks 5 and 8
Description: • The proportion of patients in each treatment group who were Responders at Week 2 and who continued to be Responders at Weeks 5 and 8.
Time Frame: Prospective
Population: Intent to Treat Population
Measure: Number; unit: participants
Arm/Group | hCRF | Placebo
Number analyzed (Participants) | 100 | 100
participants
  Week 2 | 78 | 62
  Week 5 | 62 | 48
  Week 8 | 57 | 42

4. Secondary Outcome: Change From Baseline in the 10-Item Neurological Examination Score at Weeks 2, 5, 8 12 and 16 (or Early Discontinuation)
Description: Change from Baseline in the 10-Item Neurological Examination Score at Weeks 2, 5, 8, 12 (or Early Study Drug Discontinuation), and 16 (or 4-week follow-up visit). Each item is scored from 0 (normal) to 4 (severely abnormal) except for speech (0-3) for a total range of 0-39. Total score for each patient was the sum of each item score. Change is calculated as the follow-up score minus the baseline score; a negative value indicates improvement.
Time Frame: Prospective
Population: Intent to Treat population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | hCRF | Placebo
Number analyzed (Participants) | 100 | 100
Scores on a scale
  Week 2 | -0.1 (2.3) | -0.1 (2.7)
  Week 5 | 0.2 (2.9) | 0.4 (3.0)
  Week 8 | 0.3 (3.1) | 0.5 (3.3)
  Week 12 | 0.1 (3.1) | 0.7 (3.4)
  Last Visit | 0.1 (3.1) | 0.8 (3.4)

5. Secondary Outcome: Change From Baseline in the Karnofsky Performance Score
Description: Change from Baseline in the Karnofsky Performance Score at Weeks 2, 5, 8, 12 and 16.The Karnofsky score runs from 100 to 0, where 100 is "perfect" health and 0 is death. Although practitioners occasionally assign performance scores in between standard intervals of 10 as follows:
  100 - Normal; no complaints; no evidence of disease. 90 - Able to carry on normal activity; minor signs or symptoms of disease. 80 - Normal activity with effort; some signs or symptoms of disease. 70 - Cares for self; unable to carry on normal activity or to do active work. 60 - Requires occasional assistance, but is able to care for most of his personal needs.
  50 - Requires considerable assistance and frequent medical care. 40 - Disabled; requires special care and assistance. 30 - Severely disabled; hospital admission is indicated although death not imminent.
  20 - Very sick; hospital admission necessary; active supportive treatment nec
Time Frame: Prospective
Population: Intent to Treat population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | hCRF | Placebo
Number analyzed (Participants) | 100 | 100
Scores on a scale
  Week 2 | -0.5 (7.4) | -2.2 (8.5)
  Week 5 | -2.1 (9.6) | -2.6 (8.8)
  Week 8 | -3.2 (10.3) | -3.2 (9.0)
  Week 12 | -3.4 (10.1) | -3.3 (10.1)
  Last Visit | -3.5 (10.1) | -3.6 (10.2)

6. Secondary Outcome: Change From Baseline in the FACT-Br Quality of Life Results
Description: The FACT-Br Quality of Life Questionnaire was self-administered at Baseline, Weeks 5 and 12 (or upon Early SDD), and at the post-treatment 4-week follow-up visit (Week 16 and/or any unscheduled 4-week Follow-up).FACT-Br is a reliable and valid 50-item measure that includes FACT-G (27 items) and a brain subscale (23 items) to assess health-related quality of life in brain tumor patients. Each inventory question is scored from 0 (worst possible QOL) to 4 (best possible QOL)
Time Frame: Prospective
Population: Intent to Treat; LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | hCRF | Placebo
Number analyzed (Participants) | 75 | 71
Scores on a scale
  Week 5 | 0.6 (17.5) | -2.2 (15.8)
  Week 12 | -1.8 (20.3) | -1.9 (20.3)
  Week 16 | 01.7 (20.9) | -5.9 (20.9)

7. Secondary Outcome: Change From Baseline in Myopathy Assessment Results at Week 12 (or Early Study Drug Discontinuation) and Week 16 (or 4-week Follow-up Visit)
Description: Myopathy, using Kendall Myopathy Scale, was assessed at Baseline, Week 12 (or upon Early SDD), and at the post-treatment 4-week follow-up visit (Week 16 and/or any unscheduled 4-week Follow-up). The Kendall Myopathy Scale is a 10 point scale where 10 represents holding test position against strong pressure (best) and 0 represents no contraction palpable (worst).
Time Frame: Prospective
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | hCRF | Placebo
Number analyzed (Participants) | 78 | 77
Scores on a scale
  Week 12 | 0.1 (2.8) | -0.2 (2.2)
  Week 16 | 0.0 (2.7) | -0.3 (2.5)

8. Secondary Outcome: Maximum Percent Reduction in Dexamethasone Usage Relative to Baseline Achieved During the Study
Description: The maximum reduction in dexamethasone usage at any time during the study. Dexamethasone dosage was assessed at Weeks 0, 2, 5, 8, 12 and 16.
Time Frame: Prospective
Population: Intent to Treat population; baseline observation carried forward
Measure: Mean (Standard Deviation); unit: Percent dexamethasone dose reduction
Arm/Group | hCRF | Placebo
Number analyzed (Participants) | 95 | 92
Percent dexamethasone dose reduction | -62.7 (21.8) | -51.4 (21.5)

9. Secondary Outcome: Number of Patients Who Discontinued Study Drug Prior to the End of Week 5
Description: Numbers of patients who discontinued prior to the Week 5 assessment
Time Frame: Prospective
Population: Intent to Treat population
Measure: Number; unit: participants
Arm/Group | hCRF | Placebo
Number analyzed (Participants) | 100 | 100
participants | 29 | 39

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) were reported at each visit to Week 16
Description: Treatment-emergent adverse events (TEAEs) excluded steroid-related conditions noted on the medical history. One patient was randomized to placebo but was administered hCRF instead. For the assessment of safety, the patient data has been included based on the treatment administered rather than that originally randomized.
Arm/Group | hCRF | Placebo
Serious Adverse Events (participants affected / at risk) | 46/101 | 40/99
Other Adverse Events (participants affected / at risk) | 99/101 | 97/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | hCRF (N=101) | Placebo (N=99)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Blindness (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Brain abscess (Infections and infestations) | 1 (1) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 2 (2) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 2 (2)
Respiratory Tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Radiation injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Large cell carcinoma respiratory tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (15) | 19 (19)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 3 (3)
Convulsion (Nervous system disorders) | 7 (7) | 5 (5)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral schaemia (Nervous system disorders) | 0 (0) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 1 (1)
Hemiparesis (Nervous system disorders) | 2 (2) | 0 (0)
Intracranial hypotension (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 2 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | hCRF (N=101) | Placebo (N=99)
Flushing (Vascular disorders) | 29 (29) | 28 (28)
Headache (Nervous system disorders) | 28 (28) | 28 (28)
Injection site erythema (General disorders) | 28 (28) | 1 (1)
Oedema peripheral (General disorders) | 25 (25) | 21 (21)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 22 (22) | 21 (21)
Fatigue (General disorders) | 18 (18) | 29 (29)
Nausea (Gastrointestinal disorders) | 18 (18) | 12 (12)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 16 (16) | 11 (11)
Convulsion (Nervous system disorders) | 14 (14) | 18 (18)
Injection site reaction (General disorders) | 14 (14) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 12 (12) | 9 (9)
Diarrhoea (Gastrointestinal disorders) | 12 (12) | 4 (4)
Hemiparesis (Nervous system disorders) | 11 (11) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (10) | 9 (9)
Insmnia (Psychiatric disorders) | 9 (9) | 11 (11)
Vomiting (Gastrointestinal disorders) | 9 (9) | 9 (9)
myopathy (Musculoskeletal and connective tissue disorders) | 9 (9) | 7 (7)
Confusional state (Psychiatric disorders) | 8 (8) | 11 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 8 (8)
Gait disturbance (General disorders) | 8 (8) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 1 (1)
Vision blurred (Eye disorders) | 6 (6) | 7 (7)
Weight increased (Investigations) | 6 (6) | 7 (7)
Contusion (Injury, poisoning and procedural complications) | 6 (6) | 6 (6)
Urinary tract infection (Infections and infestations) | 6 (6) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 6 (6) | 2 (2)
Tremor (Nervous system disorders) | 6 (6) | 2 (2)
Depression (Psychiatric disorders) | 5 (5) | 10 (10)
Dizziness (Nervous system disorders) | 5 (5) | 9 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (5) | 3 (3)
Pneumonia (Infections and infestations) | 5 (5) | 3 (3)
Hypertension (Vascular disorders) | 5 (5) | 3 (3)
Oral candidiasis (Infections and infestations) | 5 (5) | 0 (0)
Diplopia (Eye disorders) | 4 (4) | 5 (5)
Balance disorder (Nervous system disorders) | 4 (4) | 5 (5)
Aphasia (Nervous system disorders) | 3 (3) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7)
Partial seizures (Nervous system disorders) | 3 (3) | 7 (7)
Ataxia (Nervous system disorders) | 3 (3) | 6 (6)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6)
Somnolence (Nervous system disorders) | 3 (3) | 5 (5)
Cushingoid (Endocrine disorders) | 2 (2) | 13 (13)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 6 (6)
Pyrexia (General disorders) | 2 (2) | 5 (5)
Brain oedema (Nervous system disorders) | 2 (2) | 5 (5)
Candidiasis (Infections and infestations) | 1 (1) | 6 (6)
Cognitive disorder (Nervous system disorders) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less